CLINICAL TRIAL: NCT01830725
Title: Relationship of Purine Metabolism Enzyme Single-Nucleotide Polymorphisms to Uric Acid Production and Response to Xanthine Oxidase Inhibitors
Brief Title: Purine Metabolism Enzyme SNP to Uric Acid Production
Status: Completed | Type: Observational
Sponsor: Keesler Air Force Base Medical Center (U.S. Federal Agency)
Collaborators: United States Air Force (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: FKE20120020H
Record Dates: First submitted 2013-04-05; First posted 2013-04-12 (Estimated); Last update posted 2016-08-30 (Estimated); Status verified 2016-08

CONDITIONS: Gout; Hyperuricemia
Keywords: Xanthine Oxidase; Gout; Hyperuricemia; SNP; Single Nucleotide Polymorphisms
MeSH Terms: conditions — Gout; Hyperuricemia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — DNA will be banked for future studies as allowed by patient consent
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Gout/Hyperuricemia: Subjects with a diagnosis of hyperuricemia (defined as a uric acid of > 7.2 mg/dl) and/or gout.
- Control: Approximate age and gender matched controls without hyperuricemia or gout

SUMMARY:
Determine whether a relationship exists between polymorphisms of the genes XDH, HPRT1, and PRPS1 and gout, hyperuricemia, or the dose of xanthine oxidase (XO) inhibitors to reach a goal serum uric acid of less than 6 mg/dL. This study is observational in nature as no dose adjustment of XO inhibitors will be made by study investigators.

DETAILED DESCRIPTION:
Background: Our recent gout study demonstrated a relationship between the xanthine oxidase (XO) single nucleotide polymorphism (SNP) 2107A>G to the dose of allopurinol needed to reach a goal serum uric acid level of 6 mg/dL or less. This study had some limitations but suggests that specific SNPs could be related to dose of allopurinol needed to treat.

Objective: To determine the relationship of multiple purine enzyme SNPs of genes encoding PRPS1, HPRT1, and XO to the dose of xanthine oxidase inhibitor needed to achieve a goal treatment uric acid level of less than 6 mg/dL. Another primary outcome will be to determine relationship of two XO SNPs to hyperuricemia/gout. A secondary outcome will be to determine the frequency of these SNPs tested.

Design: Patients will be consented for enrollment in either the gout/hyperuricemia group or a control group. Control group patients will have neither gout nor hyperuricemia. No patients will be enrolled if they are overproducers of uric acid. It is anticipated that 200 patients will be enrolled in each group for a total of 400 patients over the next 2 years.

ELIGIBILITY:
Inclusion Criteria:

* The study will be open to all adults over age 18 years of age who satisfy at least one of the conditions below:
* Have asymptomatic hyperuricemia (serum uric acid level > 7.0 mg/dL) on at least 2 separate occasions,
* Clinical diagnosis of gout,
* Have neither asymptomatic hyperuricemia or gout but will serve as part of the control group (approximate age/gender matched control)

Exclusion Criteria:

* To best isolate the relationship between purine enzyme SNPs to hyperuricemia or gout and its treatment, factors which could elevate the serum uric acid level independent of protein function need to be excluded. Specifically, patients who are "overproducers" of serum uric acid will be excluded:
* Have a myeloproliferative disorder (hematologic malignancy such as leukemia or lymphoma)
* Are actively receiving therapy for any neoplasia (aside from non-melanoma skin cacner)
* Have greater than 5% of skin involvement from psoriasis
* Have a known history of xanthinuria
* Consume more than 14 drinks per week of alcoholic beverages

Patients that are pregnant or nursing will not be enrolled. Patients to be enrolled in the control group will also be excluded from enrollment if they have any of the conditions above.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients for either the gout/hyperuricemia group or the control group will be recruited at the time of their evaluation in either the Internal Medicine (IM) Clinic or IM Specialties Clinic.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2012-12; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Relationship of SNPs to gout, hyperuricemia, and dose of xanthine oxidase inhibitor needed to reach goal serum uric acid level of < 6 mg/dL. | 2 years
  This study will test the relationship of 2107A>G XO to the dose of allopurinol needed to achieve a treatment goal of less than 6 mg/dL. It will also test whether or not SNPs affecting the gene for hypoxanthine phosphoribosyltransferase 1 (HPRT1) are related to gout, hyperuricemia, or the dose of XO inhibitor needed to reach a goal of 6 mg/dL. Relationships will be determined using typical non-parametric or parametric tests depending on the skew and skedasticity.
  - Determine the relationship of several SNPs in genes encoding HPRT1 and one XO SNP (2107A>G) to the dose of xanthine oxidase inhibitor needed to achieve a goal treatment uric acid level of less than 6 mg/dL.

SECONDARY OUTCOMES:
Determine frequency of SNPs tested | 2 years
  (1) Measure minor allele frequency of all SNPs tested as the number of heterozygotes present in the population recruited divided by the total number of patients recruited.

OTHER OUTCOMES:
Determine relationship of XO SNP 2107A>G and several HPRT1 SNPs to hyperuricemia/gout. | 2 years
  This study will test the relationship of 2107A>G XO to the dose of allopurinol needed to achieve a treatment goal of less than 6 mg/dL. It will also test whether or not SNPs affecting the gene for hypoxanthine phosphoribosyltransferase 1 (HPRT1) are related to gout, hyperuricemia, or the dose of XO inhibitor needed to reach a goal of 6 mg/dL. Relationships will be determined using typical non-parametric or parametric tests depending on the skew and skedasticity.
  - Determine relationship of XO SNP 2107A>G and several HPRT1 SNPs to hyperuricemia/gout.

CONTACTS AND LOCATIONS:
Overall Officials: Matthew B Carroll, MD, Principal Investigator — Keesler Medical Center
Locations (1):
- Keesler Medical Center, Keesler Air Force Base, Mississippi, United States